CLINICAL TRIAL: NCT00462072
Title: Microarray Analysis of Peripheral Blood and Tissues of Patients With Immune Mediated Inflammatory Diseases
Brief Title: Centocor Microarray Study of Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine Allergy, Immunology & Rheumatology Division, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-01
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Psoriasis; Crohn's Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Psoriasis; Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab — Subjects will be on a stable dose of methotrexate 12.5 to 20 mg per week and will be started on infliximab 5 mg/kg.

SUMMARY:
Specific Aim 1. To determine the transcriptome of peripheral blood mononuclear cells isolated monocytes and target tissues in IMIDs.

Specific Aim 2. To analyze the change in gene expression profiles in patients with Crohn's disease, psoriatic and rheumatoid arthritis before and after infliximab therapy.

DETAILED DESCRIPTION:
Our hypothesis is that hematopoietic stem cells are very sensitive to elevated levels of TNFa, which potentiates their differentiation into myeloid effector cells. During their migration from the bone marrow to the end organ, these cells express a unique set of genes that function to prime these cells to respond to critical differentiation signals. Elucidation of this transcriptome through microarray analysis will provide insight into novel drug targets and a formal understanding of the biochemical and molecular genetic events linking IMIDs. To test our hypothesis, will determine the transcriptome in peripheral blood mononuclear cells and isolated monocytes from 20 normal healthy donors, 10 patients with psoriatic arthritis, 10 patients with psoriasis, 10 patients with Crohn's disease and 10 patients with rheumatoid arthritis. The transcriptome will also be examined in inflamed intestinal tissue from patients with Crohn's disease, psoriatic skin and synovial tissue from patients with rheumatoid and psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

Rheumatoid Arthritis

* 18 years of age or older
* 3 years duration of disease or less
* Must meet ACR criteria
* 3 tender or swollen joints
* Positive RF or anti-CCP antibodies or evidence of erosions on plain radiographs
* CRP > 1.5
* Non-responder to methotrexate, but on a stable dose of 12.5 to 20 mg/week
* Only subjects scheduled to receive infliximab as part of their care are eligible to participate.

Crohn's disease

* 12 years of age or older
* Clinical and endoscopic confirmation of disease
* CDAI > 220 or evidence of intestinal inflammation on endoscopy
* Documented failure to conventional therapy.
* Only subjects scheduled to receive infliximab as part of their care are eligible to participate.

Psoriatic arthritis

* 18 years of age or older
* Must meet CASPAR® criteria for diagnosis
* RF and anti-CCP negative
* 3 tender or swollen joints
* Non-responder to methotrexate, but on a stable dose of 12.5 to 20 mg/week
* Only subjects scheduled to receive infliximab as part of their care are eligible to participate.

Psoriasis

* 18 years of age or older
* Total BSA > 5%

Exclusion Criteria:

* Candidates for whom the procedures would be medically contraindicated would be excluded.
* Patients with any active infections (viral or bacterial) will not be considered for inclusion into the trial.
* Patients with history of chronic infection such as hepatitis, pneumonia or chronic pyelonephritis; those with current signs or symptoms of severe or progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease including demyelinating disease such as multiple sclerosis.
* Those with history of lymphoproliferative disease such as lymphoma or signs suggestive of lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, supraclavicular, epitrochlear, or periaortic areas), or splenomegaly will be excluded.
* Patients with concomitant diagnosis of CHF, including medically controlled asymptomatic patients will not be eligible to participate.
* Any current known malignancy or history of malignancy in the last 10 years will be excluded. History of basal cell carcinoma is not excluded.
* Those with known bacterial, tuberculosis or opportunistic infections including but not limited to evidence of active cytomegalovirus , active Pneumocystis carinii, aspergillosis, or atypical mycobacterium infection within the previous 6 months will be ineligible.
* Those with known infection with Human immunodeficiency virus (HIV) or known active hepatitis B or C (including associated active hepatitis) will be excluded.
* Known substance abuse (drug or alcohol) within the previous 3 years.
* Patients who have previously taken anti-TNF therapy are not eligible.
* Patients who have been treated with DMARDS, biologic or investigational agents must wash out for at least 6 weeks prior to enrollment with the exception of those on methotrexate, who must be on a stable dose at least 2 weeks prior to start of study.
* Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening.
* Have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening.
* Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including TB.
* Have had a nontuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, Pneumocystis carinii, aspergillosis) within 6 months prior to screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 subjects were enrolled from our clinic between April 4th, 2007 and June 8th, 2009.
Pre-assignment Details: Subjects were enrolled based on protocol inclusion / exclusion criteria. Subjects were required to be starting Infliximab as a requirement for entry into the study.
Groups:
- Psoriasis (Ps): Ps subjects taking Infliximab as part of their standard of care.
- Psoriatic Arthritis (PsA): PsA subjects taking Infliximab as part of their standard of care.
- Rheumatoid Arthritis (RA): RA subjects taking Infliximab as part of their standard of care.
Period: Baseline (Week 0)
Arm/Group | Psoriasis (Ps) | Psoriatic Arthritis (PsA) | Rheumatoid Arthritis (RA)
Started | 10 | 12 | 9
Completed | 10 | 12 | 9
Not Completed | 0 | 0 | 0
Period: Week 10
Arm/Group | Psoriasis (Ps) | Psoriatic Arthritis (PsA) | Rheumatoid Arthritis (RA)
Started | 10 | 12 | 9
Completed | 10 | 12 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rheumatoid Arthritis (RA): RA subject starting Infliximab
- Psoriatic Arthritis (PsA): PsA subjects starting Infliximab
- Psoriasis (Ps): Ps subjects starting Infliximab
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Psoriasis (Ps) | Total
Number analyzed (Participants) | 9 | 12 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 10 | 27
  >=65 years | 1 | 3 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 53 (13) | 41 (15) | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 20
  Male | 1 | 6 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Baseline (Wk 0) Disease Activity Score (DAS28)
Description: The DAS28 for RA and PsA subjects is an outcome measure used in determining the severity of an individual's disease. This score is used to assess disease activity and to make and monitor treatment decisions. The baseline DAS28 is an average of the study populations baseline disease activity score prior to the administration of Infliximab (remicade). A DAS28 score of higher than 5.1 is indicative of high disease activity, whereas a DAS28 below 3.2 indicates low disease activity. A subject is considered to be in remission if they have a DAS28 lower than 2.6.
Time Frame: Baseline (Wk 0)
Population: Participant data analyzed per protocol using the following DAS28 formula [(=0.56*SQRT(Tender Joint Count)+0.28*SQRT(Swollen Joint Count)+0.36*LN(CRP(mg/L)+1)+0.014*(Visual Analogue Scale+0.96 ]
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Psoriatic Arthritis (PsA): PsA subjects starting Infliximab as part of their standard of care.
- Rheumatoid Arthritis (RA): RA subjects starting Infliximab as part of their standard of care.
Arm/Group | Psoriatic Arthritis (PsA) | Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 12 | 9
Score | 4.54 (1.24) | 6.03 (1.16)

2. Primary Outcome: Week 10 Disease Activity Score (DAS28)
Description: The DAS28 for RA and PsA subjects is an outcome measure used in determining the severity of an individual's disease. This score is used to assess disease activity and to make and monitor treatment decisions. The week 10 DAS28 is an average of the study population's week 10 disease activity score after taking infliximab (remicade) for 10 weeks. A DAS28 score of higher than 5.1 is indicative of high disease activity, whereas a DAS28 below 3.2 indicates low disease activity. A subject is considered to be in remission if they have a DAS28 lower than 2.6.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Psoriariatic Arthritis (PsA): PsA subjects taking Infliximab as part of their standard of care.
Arm/Group | Psoriariatic Arthritis (PsA) | Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 12 | 9
Score | 3.34 (1.06) | 4.13 (1.28)

3. Primary Outcome: Disease Activity Score (DAS28) Delta
Description: The DAS28 Delta for RA and PsA subjects is measure used to determine the change in the severity of an individual's disease with positive delta indicating an improvement in the severity of subject's disease and a negative delta indicating a worsening of a subject's disease. The delta score is used to monitor treatment. The week 10 DAS28 Delta is determined by calculating the average change between the wk 0 and wk 10 DAS28.
Time Frame: Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score Delta
Groups:
- Rheumatoid Arthritis: RA subjects taking Infliximab as part of their standard of care.
Arm/Group | Psoriatic Arthritis (PsA) | Rheumatoid Arthritis
Number analyzed (Participants) | 12 | 9
Score Delta | 1.21 (0.60) | 1.90 (1.48)

4. Primary Outcome: Baseline (Wk 0) Psoriasis Area and Severity Index (PASI)
Description: A PASI score for Ps subjects is an outcome measure used in determining the severity of an individual's disease. This score is used to assess disease activity and to make and monitor treatment decisions. The baseline PASI is an average of the study populations baseline disease activity score prior to the administration of infliximab (remicade). While higher PASI scores indicate more severe psoriasis, it is difficult for subjects or doctors to describe the clinical severity for any specific PASI number.
Time Frame: Baseline (Wk 0)
Population: PASI formula PASI = 0.1 * (erythemahead + indurationhead + desquamationhead) * Area Scorehead + 0.2 * (erythemaarm + indurationarm + desquamationarm) * Area Scorearm + 0.3 * (erythematorso + indurationtorso + desquamationtorso) * Area Scoretorso + 0.4 * (erythemaleg + indurationleg + desquamationleg) * Area Scoreleg
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Psoriasis (Ps)
Number analyzed (Participants) | 10
Index | 5.26 (1.82)

5. Primary Outcome: Baseline (Wk 10) Psoriasis Area and Severity Index (PASI)
Description: A PASI score for Ps subjects is an outcome measure used in determining the severity of an individual's disease. This score is used to assess disease activity and to make and monitor treatment decisions. The week 10 PASI is an average of the study population's week 10 disease activity score after taking infliximab (remicade) for 10 weeks.
Time Frame: Week 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Psoriasis (Ps)
Number analyzed (Participants) | 10
Index | 2.31 (5.85)

6. Primary Outcome: Psoriasis Area and Severity Index (PASI) Delta
Description: The PASI Delta for Ps subjects is a measure used to determine the change in the severity of an individual's disease with a positive delta indicating an improvement in the severity of subject's disease and a negative delta indicating a worsening of a subject's disease. The delta score is used to monitor treatment. The week 10 PASI Delta is determined by calculating the average change between the wk 0 and wk 10 PASI.
Time Frame: Week 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Index Delta
Arm/Group | Psoriasis (Ps)
Number analyzed (Participants) | 10
Index Delta | 2.95 (5.42)

ADVERSE EVENTS:
Arm/Group | Psoriasis (Ps) | Psoriatic Arthritis (PsA) | Rheumatoid Arthritis (RA)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No